CLINICAL TRIAL: NCT06096558
Title: Effects of Melatonin, as a Dietary Supplement, on Glycemic Parameters, Cardiovascular Disease Risk Factors, Bone Metabolism Markers and Quality of Life in Peritoneal Dialysis Patients
Brief Title: The Effects of Melatonin on Cardiovascular and Bone Metabolism Markers in Peritoneal Dialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, zahra yari, assistant professor, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1402.034
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Peritoneal Dialysis
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Active Comparator)
  Interventions: Dietary Supplement: Melatonin
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — 5 mg Melatonin in one tablet, 30 minutes before night sleep
  Arms: Melatonin
Other: placebo — 1 tablet of placebo (starch)
  Arms: placebo

SUMMARY:
The aim of this double-blind randomized clinical trial is to determine the effects of Melatonin on cardiovascular disease risk factors, bone metabolism markers, serum concentrations of advanced glycated end products and quality of life in peritoneal dialysis patients. Forty patients from peritoneal dialysis centers will randomly assign to either Melatonin or placebo group. The patients in Melatonin group will receive 5 mg Melatonin (as 1 tablet) daily for 10 weeks, while the placebo group will receive identical placebo. At the baseline and the end of the study,7 ml blood will be collected from each patient after a 12-14-hours fasting and Serum concentrations of malondialdehyde; high sensitivity c-reactive protein; Soluble intercellular adhesion molecule-1; glucose; pentosidine; carboxy-methyl lysine; Procollagen 1 Intact N-Terminal Propeptide; Tartrate-resistant acid phosphatase 5b; osteoprotegerin; Receptor activator of nuclear factor kappa-Β ligand; Intact parathyroid hormone; triglyceride; total cholesterol; High-density lipoprotein cholesterol; low-density lipoprotein cholesterol; lipoprotein-a; albumin; calcium; phosphorous; and also systolic blood pressure; diastolic blood pressure and questionnaires including quality of life; quality of sleep and depression will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Continuous Ambulatory Peritoneal Dialysis for 6 months or more
* Body mass index (BMI) below 35

Exclusion Criteria:

* Infectious diseases (especially peritonitis) and inflammatory diseases Liver diseases
* Past medical history of cancer Receiving glucocorticoid drugs, non-steroidal anti-inflammatory drugs
* Receiving Melatonin supplements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Lp (a) | 10 weeks
  Serum concentrations of lipoprotein-a
MDA | 10 weeks
  Serum concentrations of malondialdehyde
hs-CRP | 10 weeks
  Serum concentrations of high sensitivity c-reactive protein
sICAM-1 | 10 weeks
  Serum concentrations of Soluble intercellular adhesion molecule-1
glucose | 10 weeks
  serum concentration of fasting glucose
pentosidine | 10 weeks
  serum concentration of pentosidine
carboxy-methyl lysine | 10 weeks
  serum concentration of carboxy-methyl lysine
P1NP | 10 weeks
  serum concentration of Procollagen 1 Intact N-Terminal Propeptide
Osteoprotegerin | 10 weeks
  Serum concentrations of Osteoprotegerin
TRACP5b | 10 weeks
  Serum concentrations of Tartrate-resistant acid phosphatase 5b
RANKL | 10 weeks
  Serum concentrations of Receptor activator of nuclear factor kappa-Β ligand
Systolic blood pressure | 10 weeks
  Systolic blood pressure (mmHg)
Diastolic blood pressure | 10 weeks
  Diastolic blood pressure (mmHg)
triglyceride | 10 weeks
  Serum concentrations of triglyceride
Total cholesterol | 10 weeks
  Serum concentrations of total cholesterol
HDL-C | 10 weeks
  Serum concentrations of High-density lipoprotein cholesterol
LDL-C | 10 weeks
  Serum concentrations of low-density lipoprotein cholesterol
Quality of life index (KDQOL) questionnaire | 10 weeks
  Filling the kidney disease quality of life index (KDQOL) questionnaire
the Beck depression test | 10 weeks
  Filling the Beck depression test
Quality of sleep Pittsburgh Sleep Quality Index (PSQI) questionnaire | 10 weeks
  Filling the Pittsburgh Sleep Quality Index (PSQI) questionnaire

SECONDARY OUTCOMES:
albumin | 10 weeks
  Serum concentrations of albumin
calcium | 10 weeks
  Serum concentrations of calcium
phosphorous | 10 weeks
  Serum concentrations of phosphorous
iPTH | 10 weeks
  Serum concentrations of Intact parathyroid hormone

REFERENCES:
- [Derived] Movahedian M, Tabibi H, Atabak S, Hedayati M, Najafi I, Seyrafian S, Rouhani MH. Effects of melatonin on advanced glycation end products, inflammation, and oxidative stress in peritoneal dialysis patients: a randomized controlled trial. Sci Rep. 2025 Oct 22;15(1):36896. doi: 10.1038/s41598-025-20792-2. PMID 41125682